CLINICAL TRIAL: NCT00060307
Title: A Phase II Study of OSI-774 (NSC-718781) in Patients With Locally Advanced or Metastatic Papillary Histology Renal Cell Cancer
Brief Title: Erlotinib in Treating Patients With Locally Advanced or Metastatic Papillary Renal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03059; S0317; U10CA032102 (NIH); CDR0000301594 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Recurrent Renal Cell Cancer; Stage III Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Erlotinib Hydrochloride

ARMS (1):
- Treatment (erlotinib hydrochloride) (Experimental): Patients receive oral erlotinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well erlotinib works in treating patients with locally advanced or metastatic papillary renal cell (kidney) cancer. Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess response (confirmed complete and partial response) of patients with locally advanced or metastatic papillary histology renal cell cancer treated with OSI-774.

II. To assess the overall survival and 6-month probability of treatment failure of this group of patients.

III. To evaluate the qualitative and quantitative toxicities of this regimen. IV. To investigate in a preliminary manner the association of tumor response with tumor expression of epidermal growth factor receptor and status of von Hippel Lindau gene mutation.

OUTLINE:

Patients receive oral erlotinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 5-20 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed papillary histology renal cell carcinoma which is metastatic (M1); patients with unresectable primary tumor (but M0) are also eligible; patients who have undergone a prior nephrectomy should have histologic confirmation of the metastatic nature of at least one distant site of disease
* Patients must have available and be willing to submit representative slides for central pathology review; these must be sent within 28 days of registration; failure to submit these materials will make the patient ineligible for this study
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension; soft tissue disease that has been radiated in the 2 months prior to registration is not assessable as measurable disease; soft tissue disease within a prior radiation field that was radiated greater than 2 months prior to registration must have progressed to be considered assessable, and patients also must have measurable disease outside of the irradiated field; X-rays, scans or physical examinations used for tumor measurement must have been completed within 28 days prior to registration; X-rays, scans or physical examinations for non-measurable disease must have been completed within 42 days prior to registration
* Patients with metastatic disease who have a resectable primary tumor and are deemed a surgical candidate may have undergone resection and have recovered from surgery; at least 28 days must have elapsed since surgery and patient must have recovered from any adverse effects of surgery
* Patients with a history of brain metastases or who currently have treated or untreated brain metastases are not eligible; patients with clinical evidence of brain metastases must have a brain CT or MRI negative for metastatic disease within 56 days prior to registration
* Patients must have available and be willing to submit archived tumor tissue that will yield sixteen 5 micron unstained slides for molecular correlative studies related to the EGFR and vHL pathways
* Patients must not have received prior chemotherapy or immunotherapy
* Patients may have received prior radiation therapy, but must have measurable disease outside the radiation port; at least 21 days must have elapsed since completion of prior radiation therapy; patients must have recovered from all associated toxicities at the time of registration
* Patients must have a Zubrod performance status of 0 - 2
* WBC ≥ 3,000/μl obtained within 14 days prior to registration
* ANC ≥ 1,500/μl obtained within 14 days prior to registration
* Platelet count ≥ 100,000/μl obtained within 14 days prior to registration
* Serum bilirubin ≤ 1.5 x institutional upper limits of normal
* Serum transaminase (SGOT or SGPT) must be ≤ 1.5 x the institutional upper limit of normal unless the liver is involved with the tumor, in which case serum transaminase (SGOT or SGPT) must be ≤ 5 x the institutional upper limit of normal; these tests must be obtained within 14 days prior to registration
* Serum creatinine must be ≤ 2 X the institutional upper limit of normal
* Patients with a known history of the following corneal diseases are not eligible: dry eye syndrome, Sjogren's syndrome, keratoconjunctivitis sicca, exposure keratopathy, Fuch's dystrophy or other active disorders of cornea
* Patients known to be HIV-positive and receiving combination anti-retroviral therapy are not eligible due to possible pharmacokinetic interactions with OSI-774
* Patients must not have gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease; patients must either be able to swallow and/or receive enteral medications via gastrostomy feeding tube; patients with intractable nausea or vomiting are not eligible
* Pregnant or nursing women may not participate on this study because OSI-774 is an epidermal growth factor inhibitor with the potential for teratogenic or abortifacient effects based on the data suggesting that EGFR expression is important for normal organ development; there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with OSI-774; women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* If day 14, 21, 28 or 42 falls on a weekend or holiday, the limit may be extended to the next working day; in calculating days of tests and measurements, the day a test or measurement is done is considered to be day 0; therefore, if a test is done on a Monday, the Monday two weeks later would be considered day 14; this allows for efficient patient scheduling without exceeding the guidelines
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and ID number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2003-05; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Response probability (confirmed complete and partial response) | Up to 3 years

SECONDARY OUTCOMES:
Time to treatment failure | 6 months
Overall survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gordon, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group, San Antonio, Texas, United States